CLINICAL TRIAL: NCT06257836
Title: Medial Patellofemoral Ligament Reconstruction in Children - a 2-8 Years Follow-up Study
Acronym: MPFL
Status: Active, not recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, PhD, MD, Aarhus University Hospital
Other Study IDs: Danish EC: 1-10-72-299-21
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Medial Patellofemoral Dislocation; Medial Patellofemoral Ligament Reconstruction
Keywords: MPFL, Knee, Medial Patellofemoral Ligament, Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MPFL reconstruction with quadriceps graft: Children with medial patellofemoral reconstruction operated with epiphyses sparing quadriceps technique from 2016-2022.
  Interventions: Other: MPFL-reconstruction
- Healthy Cohort: A healthy cohort matched on age (+/- 2 years) and gender

INTERVENTIONS:
Other: MPFL-reconstruction — Children with patella dislocations are operated from 2016-2022 with a quadriceps knee cap stabilization technique.
  Groups: MPFL reconstruction with quadriceps graft

SUMMARY:
The purpose of this project is to investigate the treatment outcome after MPFL reconstruction in children as a treatment for chronic patellar instability, where the superficial part of the quadriceps tendon is fixed to the femur with anchors.

The outcome will be compared with a healthy cohort matched on age and gender.

DETAILED DESCRIPTION:
Lateral patella dislocation (PL) is defined as a total dislocation of the patella out of the trochlea.

In chronic patella instability, where the patella has been repeatedly dislocated, the treatment is most often surgical. The main ligamentous structure that stabilizes the patella against lateralization is the medial patello-femoral ligament (MPFL). The MPFL is a centimeter-thin ligamentous structure that runs from the upper medial patellar border to the medial femoral epicondyle. This ligament is torn in more than 90% of cases of PL and healing of the ligament is often insufficient, especially if there are predisposing factors in the knee joint such as dysplasia of the patello-femoral joint, high standing patella (patella alta) and hypermobility.

MPFL reconstruction (MPFL-r) can be performed with many different surgical techniques, but the basic principle is to use autologous tendon tissue to create a new MPFL by anchoring the new tendon tissue to the medial patellar border and the medial femoral epicondyle, while ensuring isometry of the reconstruction.

A number of different methods have been described for anchoring the new MPFL to the patella and femoral condyle.

The most commonly used type of graft for MPFL-r is the gracilis tendon, which is fixed with screws in the femur bone preceded by drilling a channel in the femoral condyle.

In non-grown patients, the growth zone of the distal femur is very close to the anatomical attachment of the MPFL. This poses a problem as a reaming that hits the growth zone carries a theoretical risk of compromising growth around the knee.

In addition, up to 50% of patients describe pain at 1 year after surgery if screw fixation is used in the medial femoral condyle.

A new MPFL-r method using a superficial portion of the quadriceps tendon fixed with an anchor provides a good 2-year result compared to gracilis tendon and screw fixation.

The effectiveness and long-term efficacy of MPFL surgery with the quadriceps tendon for children is not well described in the literature.

At the Department of Sports Traumatology in Aarhus, Denmark, the quadriceps technique has been used on non-adult patients since 2016.

In this study, the investigators want to include the 80 patients who have undergone this MPFL-r since 2016 with the quadriceps tendon technique and have a minimum of 2 years of follow-up. This patient group will compared to a healthy cohort matched on age and gender.

ELIGIBILITY:
Inclusion Criteria - Intervention group:

* MPFL-reconstruction with Quadriceps tendon graft
* Open physis at surgery date
* Minimum 2 years Follow up

Exclusion Criteria - Intervention group:

* More surgeries in index knee
* MPFL-r in opposite knee
* MPFL revision in index knee

Inclusion Criteria - Healthy group:

* No knee problems

Exclusion Criteria - Healthy group

* None
* No knee problems

Ages: 14 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients who have undergone MPFL quadriceps surgery as children in the period 2016-2022 at Aarhus University Hospital and have more than 2 years of follow-up. The patients will be 14-23 years old at the time of referral.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Kujala (Anterior Knee Pain Scale) | 24 month
  Patient reported outcome score, 0=worst and 100=best

SECONDARY OUTCOMES:
Donor site morbidity score, 0=worst and 100=best | 24 month
  Patient reported outcome score
Numerical Rating Scale (NRS-pain score) | 24 month
  Patient reported outcome score, 0=Best and 10=worst
Tegner (Activity Score) | 24 month
  Patient reported outcome score, 0=worst and 10=best
Knee pain | 24 month
  Palpatory pain in relation to graft fixation in femur on a four-point likert scale (0=no pain, 1=mild pain, 2=moderate pain, 4=severe pain)
One-legged single hop for distance | 24 month
  Physical performance test
One-legged triple hop for distance | 24 month
  Physical performance test
Side-to-side hop test | 24 month
  Physical performance test
Quadriceps Strength test | 24 month
  Physical performance test. Hand held dynamometry
Gluteus Medius Strength test | 24 month
  Physical performance test. Hand held dynamometry

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Sports Trauma, Palle Juul-Jensens Boulevard 99, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No